CLINICAL TRIAL: NCT01565005
Title: Microcephaly Genetic Deficiency in Neural Progenitors: Genotyping, Phenotyping and Functional Neuro-anatomy and Neurobiology Comparative Primitive Microcephaly (MCPH) and the Fanconi Anemia (FA)
Brief Title: Microcephaly Genetic Deficiency in Neural Progenitors
Acronym: MICROFANC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P 100128
Record Dates: First submitted 2012-02-29; First posted 2012-03-28 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Microcephaly
Keywords: MCPH; FANCONI ANEMIA
MeSH Terms: conditions — Microcephaly; Fanconi Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Microcephaly: Microcephaly Intellectual abilities Cranial MRI
- FANCONI ANEMIA

SUMMARY:
The purpose of this study is to:

I. Compare neuroradiological phenotype and cognitive functioning of MCPH patients caused by ASPM mutations already characterized and published (Passemard et al. 2009a) with other MCPH-related patients (patients with MCPH1, WDR62, CDK5RAP2, CEP 152, CENPJ, STIL, or PCNT mutations)

II. Describe the neuro-radiological and cognitive phenotype of microcephalic patients suffering from Fanconi anemia, and compared them to subjects with:

* Fanconi anemia but normal OFC (head circumference)
* MCPH patients
* Healthy control subjects Our hypothesis is that mutations in genes responsible of microcephaly impact differentially cortical brain development and functioning

DETAILED DESCRIPTION:
Phenotyping study on 2 different cohorts of rare disease affected patients:

* Group1: MCPH (including different MCPH subtypes)
* Group2: Fanconi Anemia (with or without microcephaly)

Inclusion criteria:

Common to each group:

* Age > 3 years
* Access to french "Social Security"
* No contraindication for MRI

Group1:

* Primary microcephaly without gross malformation within or extra nervous central system
* OFC < -2SD at birth and < -3 SD after age 6months
* Mutation in one MCPH gene

Group2:

Proven Fanconi Anemia with:

* Positive chromosome breakage blood test
* One of the 3 following elements:

FANCD2 positive test Fibroblast sensitivity to mitomycin Mutation in one FANC gene

Control subjects:

* No antecedent
* Normal education

Aims:

1. Description of neurological, neuropsychological and radiological phenotype for each group
2. Phenotype comparison:

   * groups 1&2
   * group1 or 2 with control subjects
   * different MCPH subtypes within group1
   * with or without microcephaly within group2
3. Epidemiological data on these rare diseases in our population

Protocol:

Patients from both groups and control subjects will be evaluated in CIC for 1 day ½. They will be examined by a child neurologist and a geneticist. All of them will have cranial MRI (1.5Tesla). Neuropsychological assessment will be performed (Wechsler scales) for patients and control subjects.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 3 years:

* Microcephalic phenotype consistent with MCPH (recruitment already done as part of a network GIS-Rare Diseases Institute). MCPH patients have already been selected in the cohort "Robert Debré."
* Holders of a Fanconi anemia characterized in terms of cytogenetics, enzyme and/or molecular (patients in the cohort "Saint Louis" followed by the KRC rare aplastic anemia)
* Healthy controls aged ≥ 5 years siblings of patients with Fanconi Anemia

Exclusion Criteria:

Patients with Fanconi anemia:

* bone marrow < 3 years
* Post-transplantation neurological complications
* developmental, genetic or environmental additional pathology

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group1:
  * Primary microcephaly without gross malformation within or extra nervous central system
  * OFC < -2SD at birth and < -3 SD after age 6months
  * Mutation in one MCPH gene
  Group2:
  Proven Fanconi Anemia with:
  * Positive chromosome breakage blood test
  * One of the 3 following elements:
  FANCD2 positive test Fibroblast sensitivity to mitomycine Mutation in one FANC gene
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Compare neuroradiological phenotype and cognitive functioning with other MCPH-related patients | 3 years
  The purpose of this study is to:
  Compare neuroradiological phenotype and cognitive functioning of MCPH patients caused by ASPM mutations already characterized and published (Passemard et al. 2009a) with other MCPH-related patients (patients with MCPH1, WDR62, CDK5RAP2, CEP 152, CENPJ, STIL, or PCNT mutations)

SECONDARY OUTCOMES:
Establish a clear organizational chart for the diagnosis of primary microcephaly | 3 years
  I. Establish a clear organizational chart for the diagnosis of primary microcephaly from the detailed description of the patient's phenotype
  II. Establish epidemiological data on the molecular genetic causes involved in human primary microcephaly

CONTACTS AND LOCATIONS:
Overall Officials: Alain VERLOES, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Parsi
Locations (1):
- Robert Debre Hospital, Paris, France

REFERENCES:
- [Derived] Gins C, Guimiot F, Drunat S, Prevost C, Rosenblatt J, Capri Y, Letard P, Khung-Savatovsky S, Mahi Henni MA, Elalaoui SC, Alison M, Guilmin Crepon S, Gressens P, Verloes A, Basto R, El Ghouzzi V, Passemard S. Radial Microbrain (Micrencephaly) Is Caused by a Recurrent Variant in the RTTN Gene. Neurol Genet. 2025 Mar 26;11(2):e200221. doi: 10.1212/NXG.0000000000200221. eCollection 2025 Apr. PMID 40151166
- [Derived] Ruaud L, Drunat S, Elmaleh-Berges M, Ernault A, Guilmin Crepon S; MCPH Consortium; El Ghouzzi V, Auvin S, Verloes A, Passemard S. Neurological outcome in WDR62 primary microcephaly. Dev Med Child Neurol. 2022 Apr;64(4):509-517. doi: 10.1111/dmcn.15060. Epub 2021 Sep 25. PMID 35726608
- [Derived] Nasser H, Vera L, Elmaleh-Berges M, Steindl K, Letard P, Teissier N, Ernault A, Guimiot F, Afenjar A, Moutard ML, Heron D, Alembik Y, Momtchilova M, Milani P, Kubis N, Pouvreau N, Zollino M, Guilmin Crepon S, Kaguelidou F, Gressens P, Verloes A, Rauch A, El Ghouzzi V, Drunat S, Passemard S. CDK5RAP2 primary microcephaly is associated with hypothalamic, retinal and cochlear developmental defects. J Med Genet. 2020 Jun;57(6):389-399. doi: 10.1136/jmedgenet-2019-106474. Epub 2020 Feb 3. PMID 32015000